CLINICAL TRIAL: NCT03622996
Title: Noncontact Vital Sign Monitoring Using Impulse Radio Ultra-wideband (IR-UWB) Radar in Neonates and Children
Brief Title: Noncontact Vital Sign Monitoring Using IR-UWB Radar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Hyun-Kyung Park, MD, PhD, Hanyang University
Other Study IDs: NRF-2017M3A9E2064735
Record Dates: First submitted 2018-07-14; First posted 2018-08-09 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: NICU

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Contact sensors can cause injuries and infections in newborn infants with fragile skin. The impulse radio ultra-wideband (IR-UWB) radar is recently demonstrated in adults as a contactless method to measure heart rate. The purpose of this study is to assess heart rate (HR) in neonates using IR-UWB radar and evaluate its accuracy, compared to the electrocardiogram (ECG) in the neonatal intensive care unit (NICU).

Methods: HR is recorded in newborn infants using both IR-UWB radar 35 cm away from the chest and ECG simultaneously in the NICU. The HR data during sleeping/calm state are automatically collected by a software algorithm. A total values averaged from a 30-second window every 10 s is used for the analysis. Data acquired on the same patient with standard electrocardiogram has been used for comparison.

DETAILED DESCRIPTION:
Vital sign is recorded by the radar and bedside ECG simultaneously in supine position within an open-air crib.

The three electrodes of the ECG are attached at the standard positions and connected to the BSM-6501K patient monitor (Nihon Kohden, Tokyo, Japan), and vital signs are recorded and extracted.

The data from the radar is connected to a computer through a USB interface, and signal processing has been automatically performed by a software algorithm described by our previous study. A Fourier transform decomposes a signal with respect to time into a frequency component.

Vital sign is recorded continuously, and digital outputs are extracted from periods when no large noise or fluctuation occurs in both methods. While vital sign acquisition is significantly interfered with moving extensively, being in nursing care, repetitive myoclonus, hiccupping, flopping, or crying, the IR-UWB radar system stops the measurements and deletes the motion-contaminated observations automatically by itself. To investigate the artifact and interference by body movement during measurement, the level of movement is integrated based on the change of distance of the body from the radar. The radar transmits dozens of these signals (frames) to the computer every second, and the frame would not be changed if there was no movement within the range of the radar. However, if there is any movement, the difference of two frames (previous - current) is calculated.

ELIGIBILITY:
Inclusion Criteria:

* full-term neonates (> 37 weeks of gestational age)

Exclusion Criteria:

* patients with congenital anomalies

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We prospectively enrolls clinically stable full-term neonates (> 37 weeks of gestational age) who do not use any respiratory support and have stable vital signs at the NICU
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate (total time of successful detection/total measurement time) between the IR-UWB radar and conventional monitor for HR and RR measurement | newborns (≥ 37 weeks gestational age) who are admitted in NICU within 28 days of birth (breathing without any respiratory/oxygen support)
  to assess the potential of IR-UWB radar for monitoring vital signs in neonates, compared to the gold standard monitoring in the NICU
Correlation by Pearson coefficient between the IR-UWB radar and conventional monitor for HR and RR measurement | newborns (≥ 37 weeks gestational age) who are admitted in NICU within 28 days of birth (breathing without any respiratory/oxygen support)
  to evaluate accuracy of IR-UWB radar for monitoring vital signs in neonates, compared to the gold standard monitoring in the NICU
Mean difference by Bland-Altman analysis between the IR-UWB radar and conventional monitor for HR and RR measurement | newborns (≥ 37 weeks gestational age) who are admitted in NICU within 28 days of birth (breathing without any respiratory/oxygen support)
  to evaluate accuracy of IR-UWB radar for monitoring vital signs in neonates, compared to the gold standard monitoring in the NICU
Signal matching (%), defined bpm difference ≤ 5, between the IR-UWB radar and conventional monitor for HR measurement | newborns (≥ 37 weeks gestational age) who are admitted in NICU within 28 days of birth (breathing without any respiratory/oxygen support)
  to evaluate accuracy of IR-UWB radar for monitoring heart rate in neonates, compared to the gold standard monitoring in the NICU

CONTACTS AND LOCATIONS:
Overall Officials: JH Ahn, Study Director — Hanyang University, Seoul, Korea
Locations (1):
- Hanyang University College of Medicine, Seoul, South Korea